CLINICAL TRIAL: NCT00603291
Title: A 52-Week, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Safety and Efficacy of Lorcaserin Hydrochloride in Overweight and Obese Patients With Type 2 Diabetes Mellitus Managed With Oral Hypoglycemic Agent(s)
Brief Title: BLOOM-DM: Behavioral Modification and Lorcaserin for Overweight and Obesity Management in Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APD356-010
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-08

CONDITIONS: Obesity
Keywords: obesity; weight loss; lorcaserin; APD356; BLOOM-DM; hypertension; dyslipidemia; sleep apnea; glucose tolerance; cardiovascular disease; Arena
MeSH Terms: conditions — Obesity; Weight Loss; Hypertension; Dyslipidemias; Sleep Apnea Syndromes; Cardiovascular Diseases | interventions — lorcaserin; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lorcaserin 10 mg QD (Experimental): Lorcaserin 10 mg tablet each morning and placebo tablet each evening
  Interventions: Drug: Lorcaserin 10 mg once daily (QD)
- Lorcaserin 10 mg BID (Experimental): Lorcaserin 10 mg tablet each morning and evening
  Interventions: Drug: Lorcaserin 10 mg twice a day (BID)
- Matching Placebo (Placebo Comparator): Matching placebo tablet each morning and evening
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Lorcaserin 10 mg once daily (QD) — Lorcaserin 10 mg tablet each morning and placebo tablet each evening for a duration of 52 weeks.
  Other Names: APD356
  Arms: Lorcaserin 10 mg QD
Drug: Lorcaserin 10 mg twice a day (BID) — Lorcaserin 10 mg tablet each morning and evening for a duration of 52 weeks.
  Other Names: APD356
  Arms: Lorcaserin 10 mg BID
Drug: Matching Placebo — Matching placebo tablet each morning and evening for a duration of 52 weeks.
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to assess the weight loss effect of lorcaserin during and at the end of 1 year of treatment in overweight and obese patients with Type II diabetes mellitus treated with metformin, sulfonylurea (SFU), or either agent in combination with other oral hypoglycemic agents.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese men and women with type 2 diabetes mellitus that is managed with oral anti-hyperglycemic agent(s).
* Body mass index (BMI) 27 to 45 kg/m2, inclusive.
* Ability to complete a 1 year study

Exclusion Criteria:

* Pregnancy
* Use of insulin in any form, exenatide (Byetta) or pramlintide (Symlin) within 3 months prior to screening
* History of symptomatic heart valve disease
* Serious or unstable current or past medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arena Pharmaceuticals, Inc., San Diego, California, United States

REFERENCES:
- [Derived] Magkos F, Nikonova E, Fain R, Zhou S, Ma T, Shanahan W. Effect of lorcaserin on glycemic parameters in patients with type 2 diabetes mellitus. Obesity (Silver Spring). 2017 May;25(5):842-849. doi: 10.1002/oby.21798. Epub 2017 Mar 27. PMID 28345809
- [Derived] Weissman NJ, Smith SR, Fain R, Hall N, Shanahan WR. Effects of lorcaserin on pre-existing valvulopathy: A pooled analysis of phase 3 trials. Obesity (Silver Spring). 2017 Jan;25(1):39-44. doi: 10.1002/oby.21695. Epub 2016 Nov 26. PMID 27888609
- [Derived] Handelsman Y, Fain R, Wang Z, Li X, Fujioka K, Shanahan W. Lorcaserin treatment allows for decreased number needed to treat for weight and glycemic parameters in week 12 responders with >/=5% weight loss. Postgrad Med. 2016 Nov;128(8):740-746. doi: 10.1080/00325481.2016.1240591. Epub 2016 Oct 19. PMID 27659698
- [Derived] Pi-Sunyer X, Shanahan W, Fain R, Ma T, Garvey WT. Impact of lorcaserin on glycemic control in overweight and obese patients with type 2 diabetes: analysis of week 52 responders and nonresponders. Postgrad Med. 2016 Aug;128(6):591-7. doi: 10.1080/00325481.2016.1208618. Epub 2016 Jul 18. PMID 27389084
- [Derived] Nguyen CT, Zhou S, Shanahan W, Fain R. Lorcaserin in Obese and Overweight Patients Taking Prohibited Serotonergic Agents: A Retrospective Analysis. Clin Ther. 2016 Jun;38(6):1498-1509. doi: 10.1016/j.clinthera.2016.04.004. Epub 2016 May 17. PMID 27206567
- [Derived] Weissman NJ, Sanchez M, Koch GG, Smith SR, Shanahan WR, Anderson CM. Echocardiographic assessment of cardiac valvular regurgitation with lorcaserin from analysis of 3 phase 3 clinical trials. Circ Cardiovasc Imaging. 2013 Jul;6(4):560-7. doi: 10.1161/CIRCIMAGING.112.000128. Epub 2013 May 9. PMID 23661689
- [Derived] O'Neil PM, Smith SR, Weissman NJ, Fidler MC, Sanchez M, Zhang J, Raether B, Anderson CM, Shanahan WR. Randomized placebo-controlled clinical trial of lorcaserin for weight loss in type 2 diabetes mellitus: the BLOOM-DM study. Obesity (Silver Spring). 2012 Jul;20(7):1426-36. doi: 10.1038/oby.2012.66. Epub 2012 Mar 16. PMID 22421927
- See also: Arena Pharmaceuticals, Inc. Home Page — http://www.arenapharm.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Lorcaserin 10 mg Once Daily (QD): lorcaserin 10 mg QD tablets
- Lorcaserin 10 mg Twice a Day (BID): lorcaserin 10 mg BID tablets
- Matching Placebo: matching placebo tablets
Period: Overall Study
Arm/Group | Lorcaserin 10 mg Once Daily (QD) | Lorcaserin 10 mg Twice a Day (BID) | Matching Placebo
Started | 95 | 256 | 253
Completed | 75 | 169 | 157
Not Completed | 20 | 87 | 96

BASELINE CHARACTERISTICS:
Groups:
- Lorcaserin 10 mg QD: lorcaserin 10 mg QD tablets
- Lorcaserin 10 mg BID: lorcaserin 10 mg BID tablets
- Total: Total of all reporting groups
Arm/Group | Lorcaserin 10 mg QD | Lorcaserin 10 mg BID | Matching Placebo | Total
Number analyzed (Participants) | 95 | 256 | 252 | 603
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (7.98) | 53.2 (8.26) | 52.0 (9.32) | 52.7 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 137 | 137 | 327
  Male | 42 | 119 | 115 | 276

OUTCOME MEASURES:

1. Primary Outcome: Co-primary Endpoint- Percentage of Participants Achieving Greater Than or Equal to 5% Weight Loss From Baseline to Week 52
Description: The percentage of patients with a reduction from baseline body weight of 5% or more after 52 weeks.
Time Frame: Baseline and Week 52
Population: Modified Intent to Treat (MITT) with last observation carried forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Lorcaserin 10 mg BID | Lorcaserin 10 mg QD | Matching Placebo
Number analyzed (Participants) | 251 | 94 | 248
percentage of participants | 37.5 | 44.7 | 16.1
Statistical Analysis 1: Comparison: Lorcaserin 10 mg BID vs Matching Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustment for baseline body weight, baseline HbA1c stratum, and prior antihyperglycemic medication stratum; Odds Ratio (OR) = 3.14, 95% CI 2-sided [2.05 to 4.80]

2. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 52
Description: The percent change in body weight (kg) from baseline to week 52.
Time Frame: Baseline and Week 52
Population: MITT with LOCF
Measure: Least Squares Mean (Standard Error); unit: % change from baseline: body wt (kg)
Arm/Group | Lorcaserin 10 mg BID | Lorcaserin 10 mg QD | Matching Placebo
Number analyzed (Participants) | 251 | 94 | 248
% change from baseline: body wt (kg) | -4.54 (0.35) | -4.97 (0.54) | -1.48 (0.36)
Statistical Analysis 1: Comparison: Lorcaserin 10 mg BID vs Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.06, 95% CI 2-sided [-3.92 to -2.20]

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Lorcaserin 10 mg BID | Lorcaserin 10 mg QD | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 16/256 | 8/95 | 17/252
Other Adverse Events (participants affected / at risk) | 236/256 | 89/95 | 213/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin 10 mg BID (N=256) | Lorcaserin 10 mg QD (N=95) | Matching Placebo (N=252)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin 10 mg BID (N=256) | Lorcaserin 10 mg QD (N=95) | Matching Placebo (N=252)
Nausea (Gastrointestinal disorders) | 24 (26) | 8 (8) | 20 (27)
Diarrhoea (Gastrointestinal disorders) | 19 (19) | 13 (16) | 19 (23)
Constipation (Gastrointestinal disorders) | 11 (11) | 6 (8) | 12 (14)
Fatigue (General disorders) | 19 (19) | 5 (5) | 10 (11)
Upper respiratory tract infection (Infections and infestations) | 35 (46) | 19 (23) | 37 (46)
Nasopharyngitis (Infections and infestations) | 29 (37) | 22 (28) | 25 (29)
Urinary tract infection (Infections and infestations) | 23 (25) | 9 (12) | 15 (16)
Gastroenteritis viral (Infections and infestations) | 18 (19) | 5 (6) | 11 (14)
Influenza (Infections and infestations) | 15 (16) | 8 (9) | 13 (14)
Sinusitis (Infections and infestations) | 16 (18) | 5 (6) | 26 (29)
Bronchitis (Infections and infestations) | 8 (8) | 5 (6) | 11 (11)
Gastroenteritis (Infections and infestations) | 8 (8) | 5 (5) | 5 (6)
Procedural pain (Injury, poisoning and procedural complications) | 13 (13) | 0 (0) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 75 (513) | 32 (253) | 53 (321)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (15) | 10 (12) | 19 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (13) | 5 (5) | 17 (19)
Headache (Nervous system disorders) | 37 (48) | 16 (20) | 18 (24)
Dizziness (Nervous system disorders) | 18 (21) | 11 (14) | 16 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 5 (5) | 11 (11)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5) | 12 (12)
Hypertension (Vascular disorders) | 13 (14) | 6 (8) | 8 (9)
Depression (Psychiatric disorders) | 6 (6) | 5 (6) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 30 (33) | 8 (10) | 20 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No